CLINICAL TRIAL: NCT05023876
Title: Effect of Instrument Assisted Soft Tissue Mobilization in Chronic Obstructive Pulmonary Disease
Brief Title: The Effect of Instrument Assisted Soft Tissue Mobilization on Respiratory Functions in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 006
Record Dates: First submitted 2021-08-21; First posted 2021-08-27 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: COPD; Pulmonary Function; Soft Tissue Mobilization
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM group (Experimental)
  Interventions: Other: Respiratory Exercise
- Control Group (Experimental)
  Interventions: Other: IASTM+respiratory Exercise

INTERVENTIONS:
Other: IASTM+respiratory Exercise — Instrument assisted soft tissue mobilization
  Arms: Control Group
Other: Respiratory Exercise — Respiratory Exercise
  Arms: IASTM group

SUMMARY:
The aim of this study is to investigate the effect of instrument-assisted soft tissue mobilization applied to the hamstring muscle on respiratory function in patients with COPDThe patients to be included in the study will be divided into two groups by simple randomization. A group will be given breathing exercises (pursed lip breathing, diaphragmatic breathing and thoracic expansion exercises) as a home program. The other group will be given breathing exercises in the form of a home program in addition to 1 session of EDYM per week. Both groups will be evaluated before and 4 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with GOLD stage I-II COPD
* Between the ages of 40-65
* COPD in stable period
* No other respiratory disease that impairs respiratory functions such as asthma
* Knee flexion angle of 15 degrees and above in the hamstring muscle shortness test,
* Individuals without musculoskeletal problems in their lower extremities were included.

Exclusion Criteria:

* COPD patients who receive home oxygen therapy or who need oxygen therapy frequently
* COPD exacerbation, hospitalization with acute exacerbation in the last 15 days
* Pregnancy
* Kyphoscoliosis, advanced postural disorder
* Prior thoracic surgery
* Advanced heart failure
* Patients with primary pulmonary hypertension or have had a pulmonary embolism,
* Having serious neurological diseases such as Parkinson's, hemiplegia, multiple sclerosis,
* Neuromuscular disease
* Having dementia, Alzheimer's or advanced cognitive problems,
* Diagnosed with lung cancer or other malignancy,
* People with morbid obesity will not be included in the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Respiratory Function | 5 minute
  Respiratory Function evaluated with spirometer

SECONDARY OUTCOMES:
Chest circumference measurement | 5 minute
  It will be performed in a standing position with body weight evenly distributed over both lower extremities. During the tidal volume maximum inspiration and maximum expiration, the body of the person will be surrounded by a tape measure separately from the fourth intercostal space (axillary region), xiphoid process and subcostal region lines. To determine rib cage mobility, the difference between chest circumference measurements at maximum inspiration and maximum expiration will be recorded in centimeters. Measurements will be repeated for both groups before and after the application.
Popliteal angle test | 3 minutes
  Popliteal Angle Test will be used to evaluate hamstring muscle mobility. The person to be evaluated will be placed on the back with the hip and knee joints flexed to 90° and the contralateral side with the extremity extended. The person will be instructed to hold the back surface of the leg with their hands and maintain the flexion angle. Meanwhile, the inclinometer will be detected in the anterior-midline of the tibia. Then, the person will be asked to extend the knee as much as tolerated and the last degree of movement will be measured. It will be repeated before and after the application for both the treatment and control groups.
Finger-floor distance measurement | 3 minutes
  To consider the mobility of the posterior chain muscles as a whole, the finger-to-ground distance test with high reliability and sensitivity will be used. The person standing on a block with a height of 15 cm from the ground will be asked to bend forward and touch his toes without bending his knees, and at the end of the movement, the distance between the distal end of his extended fingers and the ground will be measured. Values above the block will be evaluated as minus, and values below the block will be evaluated as plus. The measurement will be repeated three times and the average value will be recorded. It will be repeated before and after the application for both the treatment and control groups.
Hand grip strength | 3 minutes
  Measurement will be taken with the patients in a sitting position, shoulder adduction, elbow flexion at 90°, forearm prono-supination neutral, and wrist joint in neutral position. 3 consecutive measurements will be provided with 60-second rest breaks between measurements and the result obtained from the average of the three measurements will be recorded. It will be repeated before and after the application for both the treatment and control groups.
6-minute walk test | 6 minute
  The 6-minute walk test (6MWT) is the most commonly used field test in patients with COPD. Participants will be asked to walk the longest distance they can walk at their own pace for a period of 6 minutes, under the supervision of a physiotherapist, in a 30-meter straight corridor. After the test is complete, the total distance walked will be recorded in meters. It will be repeated before and after the application for both the treatment and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Emine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided